CLINICAL TRIAL: NCT01448109
Title: A Randomised Blinded Placebo Controlled Trial of Hydrocortisone in Critically Ill Patients With Septic Shock
Brief Title: ADjunctive coRticosteroid trEatment iN criticAlly ilL Patients With Septic Shock
Acronym: ADRENAL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The George Institute (Other)
Collaborators: National Health and Medical Research Council, Australia (Other); Australian and New Zealand Intensive Care Society Clinical Trials Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GI-CCT372273
Record Dates: First submitted 2011-10-05; First posted 2011-10-07 (Estimated); Last update posted 2017-12-12 (Actual); Status verified 2017-09

CONDITIONS: Septic Shock
Keywords: Sepsis; Corticosteroid
MeSH Terms: conditions — Shock, Septic; Sepsis | interventions — Hydrocortisone; hydrocortisone hemisuccinate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hydrocortisone (Active Comparator)
  Interventions: Drug: Hydrocortisone
- Sterile air filled vial (Placebo Comparator)
  Interventions: Drug: Sterile air filled vial

INTERVENTIONS:
Drug: Hydrocortisone — Hydrocortisone 100mg vial (blinded) is reconstituted with 2ml of water for Injection, agitated for 20 seconds, rested for 3 minutes, contents of vial aspirated and added to 100ml bag of normal saline or 5% dextrose and given intravenously as a continuous infusion at rate of 200mg/per day for 7 days.
  Other Names: Solu-Cortef
  Arms: Hydrocortisone
Drug: Sterile air filled vial — the "sterile air filled vial" (blinded) is reconstituted with 2ml of water for Injection, agitated for 20 seconds, rested for 3 minutes, contents of vial aspirated and added to 100ml bag of normal saline or 5% dextrose and given intravenously as a continuous infusion. 2 sterile air filled vials per day for 7 days
  Arms: Sterile air filled vial

SUMMARY:
The purpose of this study is to find out whether adult patients admitted to the Intensive Care Unit with septic shock who are given hydrocortisone compared to placebo (a dummy solution), will have an improved rate of survival 90 days later.

Septic shock is the result of an infection, which triggers a complex response by the body (the inflammatory response) that causes a decrease in blood pressure and subsequently one or more organ systems to fail when blood supply to these organs is reduced. This may result in poor recovery and death. About a quarter of the people who suffer septic shock that is not rapidly reversed, will die.

When patients are admitted to Intensive Care with sepsis and/or septic shock they receive a number of therapies. These include fluids given through a drip, antibiotics, drugs to boost your blood pressure and other organ systems.

In addition to these therapies, steroids (hydrocortisone) are sometimes administered. Whether steroids are useful or not in the treatment of severe infections has been studied for more than 50 years. Previous research has suggested that the use of low dose steroid may have shortterm benefits in improving the circulation. However, there is no agreement amongst doctors around the world about whether treatment with or without low dose steroids improves the overall recovery and survival in patients with septic shock. This study would allow doctors to make informed decisions about whether the addition of low dose steroid therapy is better for patients with septic shock in intensive care.

The study will include 3800 intensive care patients who have septic shock. Each enrolled patient will be randomised to receive either Hydrocortisone 200mg or placebo daily for 7 days as a continuous intravenous infusion while in intensive care. The patient will be followed for 90 days. If the patient is discharged prior to 90 days a telephone call will be made for the followup information. At six months the patient will be contacted again for completion of a quality of life questionnaire.

DETAILED DESCRIPTION:
Primary Objective To evaluate the impact of intravenous hydrocortisone versus placebo on all cause mortality at 90 days in critically ill patients with septic shock. The hypothesis is that hydrocortisone, compared to placebo, reduces 90-day all-cause mortality in patients admitted to an ICU with septic shock. 'Shock' is defined as the need for vasopressors or inotropes to maintain a systolic blood pressure > 90 millimetres of mercury (mmHg), or mean arterial blood pressure > 60mmHg or a mean arterial pressure (MAP) target set by the treating clinician for maintaining perfusion. 'Septic shock' is shock that is secondary to sepsis

Secondary Objectives To assess the impact of intravenous hydrocortisone versus placebo on the recovery from, and the complications of, septic shock and the development of treatment related adverse reactions.

Study Design This study is a multi centre, randomised, blinded, placebo controlled trial comparing intravenous hydrocortisone with placebo in critically ill patients with septic shock.

Randomisation will be achieved via a secure interactive web based system using permuted block minimisation. Randomisation will be stratified by participating site and by operative or non-operative admission to the ICU.

The primary endpoint for this trial will be death from all causes at 90 days.

Pre defined sub groups will include the following categories:

* Operative (admitted to ICU from operating theatre or recovery room) versus non-operative admission.
* Dose of adrenaline or noradrenaline at randomisation - ≤ 15 mcg / minute versus > 15 mcg / minute.

3,800 patients will be enrolled in this study at approximately 50 - 60 study sites. Eligible patients will be randomised to receive either intravenous hydrocortisone 200mg or placebo per day for 7 days.

For all patients, data will be collected at baseline and then daily whilst the patient is in the ICU. Patients will be followed up to day 14, regardless of where the patient resides in the hospital, to monitor the development of bacteraemia. Additional follow up will occur at 90 days and at 6 months post randomisation.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or older
2. Documented site of infection, or strong suspicion of infection, with 2 of the 4 clinical signs of inflammation:

   * Core temperature > 38°C or < 35°C
   * Heart rate > 90 beats per minute
   * White cell count > 12 x 109/L or < 4 x 109/L or > 10% immature neutrophils
   * Respiratory rate > 20 breaths per minute, or PaCO2 < 32 mmHg, or mechanical ventilation.
3. Being treated with mechanical ventilation at the time of randomisation
4. Being treated with vasopressors or inotropes to maintain a systolic blood pressure > 90mmHg, or mean arterial blood pressure > 60mmHg, or a MAP target set by the treating clinician for maintaining perfusion
5. Administration of vasopressors or inotropes for = 4 hours and present at time of randomisation.

Exclusion Criteria:

1. Met all inclusion criteria more than 24 hours ago
2. Clinician expects to prescribe systemic corticosteroids for an indication other than septic shock (not including nebulised or inhaled corticosteroid)
3. Patients treated with etomidate
4. Patients receiving treatment with Amphotericin B for systemic fungal infections at time of randomisation
5. Patients with documented cerebral malaria at the time of randomisation
6. Patients with documented strongyloides infection at the time of randomisation
7. Death is deemed inevitable or imminent during this admission and either the attending physician, patient or surrogate legal decision maker is not committed to active treatment
8. Death from underlying disease is likely within 90 days
9. Patient has been previously enrolled in the ADRENAL study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3800 (Actual)
Dates: Start 2012-06-13 (Actual); Primary Completion 2017-10-22 (Actual); Study Completion 2017-11-20 (Actual)

PRIMARY OUTCOMES:
All cause mortality at 90 days after randomisation | 90 days after randomisation

SECONDARY OUTCOMES:
All-cause mortality at 28 days and 6 months after randomisation | 28 days and 6 months after randomisation
Time to resolution of shock | MAP goal for >24 hours without vasopressors or inotropes. Up to 90 days after randomisation.
  Time to resolution of shock - defined as "the time taken to achieve a clinician prescribed mean arterial pressure (MAP) goal for >24 hours without vasopressors or inotropes.
Recurrence of shock | Up to90 days after randomisation
  Recurrence of shock - defined as a new episode of shock after reversal of the initial episode.
Duration of ICU stay | Up to 90 days after randomisation
Duration of hospital stay | Up to 90 days after randomisation
Frequency and duration of mechanical ventilation | Up to 90 days after randomisation
Duration of renal replacement therapy | Up to 90 days after randomisation
Development of bacteraemia | 2 and 14 days post randomisation
Bleeding requiring blood transfusions received in the ICU | Up to 90 days after randomisation
Quality of Life assessment at 6 months. | 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Balasubramanian Venkatesh, Study Chair — The George Institute
Locations (70):
- Australia (46):
  - Blacktown Hospital, Blacktown, New South Wales
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - St Vincent's Hospital, Darlinghurst, New South Wales
  - Gosford Hospital, Gosford, New South Wales
  - St George Hospital, Kogarah, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - John Hunter Hospital, Newcastle, New South Wales
  - Nepean Hospital, Penrith, New South Wales
  - Prince of Wales Hospital, Randwick, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - The George Institute for Global Health, Sydney, New South Wales
  - Tamworth Rural Referral Hospital, Tamworth, New South Wales
  - Tweed Heads District Hospital, Tweed Heads, New South Wales
  - Calvary Mater Hospital (Newcastle), Waratah, New South Wales
  - Wollongong Hospital, Wollongong, New South Wales
  - Royal Darwin Hospital, Darwin, Northern Territory
  - Wesley Hospital, Auchenflower, Queensland
  - Prince Charles Hospital, Brisbane, Queensland
  - Mater Health Services, Brisbane, Queensland
  - Gold Coast University Hospital, Gold Coast, Queensland
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Ipswich Hospital, Ipswich, Queensland
  - Logan Hospital, Logan City, Queensland
  - Mackay Base Hospital, Mackay, Queensland
  - Nambour Hospital, Nambour, Queensland
  - Redcliffe Hospital, Redcliffe, Queensland
  - Toowoomba Hospital, Toowoomba, Queensland
  - Townsville Hospital, Townsville, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Lyell McEwin Hospital, Elizabeth Vale, South Australia
  - The Queen Elizabeth Hospital, Woodville South, South Australia
  - Royal Hobart Hospital, Hobart, Tasmania
  - Bendigo Hospital, Bendigo, Victoria
  - Monash Medical Centre, Clayton, Victoria
  - Northern Hospital, Epping, Victoria
  - St Vincent's Hospital (Melbourne), Fitzroy, Victoria
  - Footscray Hospital, Footscray, Victoria
  - Geelong Hospital (Barwon Health), Geelong, Victoria
  - Austin Hospital, Heidelberg, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
  - Sunshine Hospital, St Albans, Victoria
  - Fremantle Hospital, Fremantle, Western Australia
  - Fiona Stanley Hospital, Murdoch, Western Australia
  - Royal Perth Hospital, Perth, Western Australia
  - St John of God Hospital-Murdoch, Perth, Western Australia
- Rigshospitalet, Copenhagen, Denmark
- New Zealand (8):
  - North Shore Hospital, North Shore, Auckland
  - Waikato Hospital, Hamilton, NZ
  - Auckland City Hospital (CVICU), Auckland
  - Auckland City Hospital (DCCM), Auckland
  - Middlemore Hospital, Auckland
  - Christchurch Hospital, Christchurch
  - Tauranga Hospital, Tauranga
  - Wellington Hospital, Wellington
- Saudi Arabia (3):
  - King Abdulaziz Medical City, Riyadh
  - King Khalid University Hospital, King Saud University, Riyadh
  - King Fahad Medical City, Riyadh
- United Kingdom (12):
  - Bristol Royal Infirmary, Bristol, England
  - Ashford & St.Peter's NHS Foundation Trust, Chertsey, England
  - Queen Alexandra Hospital (Portsmouth), Cosham, England
  - Queen Elizabeth Hospital Birmingham, Edgbaston, England
  - Royal Surrey County Hospital, Guildford, England
  - Lewisham Healthcare NHS Trust, London, England
  - Guy's and St Thomas' HNS Foundation Trust, London, England
  - King's College Hospital NHS Foundation Trust, London, England
  - St Georges Healthcare NHS Trust, London, England
  - Freeman Hospital, Newcastle upon Tyne, England
  - University Hospital Southampton, Southampton, England
  - Royal Gwent Hospital, Newport, Wales

REFERENCES:
- [Derived] Daubney ER, D'Urso S, Cuellar-Partida G, Rajbhandari D, Peach E, de Guzman E, McArthur C, Rhodes A, Meyer J, Finfer S, Myburgh J, Cohen J, Schirra HJ, Venkatesh B, Evans DM. A Genome-Wide Association Study of Serum Metabolite Profiles in Septic Shock Patients. Crit Care Explor. 2024 Jan 17;6(1):e1030. doi: 10.1097/CCE.0000000000001030. eCollection 2024 Jan. PMID 38239409
- [Derived] Li W, Cornelius V, Finfer S, Venkatesh B, Billot L. Adaptive designs in critical care trials: a simulation study. BMC Med Res Methodol. 2023 Oct 18;23(1):236. doi: 10.1186/s12874-023-02049-6. PMID 37853343
- [Derived] Venkatesh B, Finfer S, Cohen J, Rajbhandari D, Arabi Y, Bellomo R, Billot L, Correa M, Glass P, Harward M, Joyce C, Li Q, McArthur C, Perner A, Rhodes A, Thompson K, Webb S, Myburgh J; ADRENAL Trial Investigators and the Australian-New Zealand Intensive Care Society Clinical Trials Group. Adjunctive Glucocorticoid Therapy in Patients with Septic Shock. N Engl J Med. 2018 Mar 1;378(9):797-808. doi: 10.1056/NEJMoa1705835. Epub 2018 Jan 19. PMID 29347874